CLINICAL TRIAL: NCT04189263
Title: IIT2018-21-Amersi-BREADS BREADS: Breast Adjuvant Diet Study
Brief Title: BREADS: Breast Adjuvant Diet Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low participant compliance, slow recruitment
Sponsor: Farin Amersi (Other)
Responsible Party: Sponsor-Investigator, Farin Amersi, Associate Professor, Surgery, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2018-21-AMERSI-BREADS
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitor; carbohydrate restricted diet
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention (Experimental): Carbohydrate restricted dietary intervention (<20 g carbohydrates/day) + standard of care aromatase inhibitors
  Interventions: Other: Carbohydrate restricted dietary intervention; Drug: standard of care aromatase inhibitors
- No dietary intervention (Active Comparator): Standard of care aromatase inhibitors
  Interventions: Drug: standard of care aromatase inhibitors

INTERVENTIONS:
Other: Carbohydrate restricted dietary intervention — Carbohydrate restricted dietary intervention (<20 g carbohydrates/day)
  Arms: Dietary intervention
Drug: standard of care aromatase inhibitors — standard of care aromatase inhibitors

SUMMARY:
This is a randomized controlled trial of a 6-month extreme carbohydrate restricted diet (20 grams total carbs/day) via phone counseling with dietitian plus aromatase inhibitor therapy vs. 6-month control with aromatase inhibitor therapy alone. Visits will occur at screening, 3 months, and 6 months. Anthropomorphic measurements (such as heart rate, weight, and body measurement) and questionnaires will be taken at all three visits. After screening, patients will be randomized to receive the carbohydrate restricted diet coaching immediately (Arm A) or to a control group (Arm B). Patients randomized to Arm A will receive weekly calls for the first 3 months of the intervention, then biweekly calls for the last 3 months of the intervention from the study dietitian. Total duration of the study is expected to be 3 years, though each patient's participation will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer
* Planning to start adjuvant hormonal therapy using an aromatase inhibitor or has started adjuvant hormonal therapy using an aromatase inhibitor
* Able to read, write, and understand English
* BMI ≥ 24 kg/m2
* Age ≥ 18 years
* ER and/or PR positive (defined as having ≥ 1% staining for ER and/or PR on IHC)
* Post-menopausal

  * The absence of menstrual cycles in women who have not undergone hysterectomy for at least 12 months preceding cancer diagnosis OR
  * History of a bilateral oophorectomy OR
  * History of a hysterectomy and age >55 OR
  * No menses for <1 year with FSh and estradiol levels in postmenopausal range according to institutional standards
* ECOG Performance Status 0 or 1
* Female
* Written informed consent obtained from subject and ability for subject to comply with requirements of the study

Exclusion Criteria:

* Use of hormonal therapy other than aromatase inhibitors
* History of other malignancy within the past 5 years, except for malignancies with a > 95% likelihood of cure (e.g. thyroid cancer, non-melanoma skin cancer)
* Already consuming a severe carbohydrate restricted (<20 g carbohydrates per day) diet or vegetarian diet
* Currently on or plans to start chemotherapy (HER2/neu targeted therapy okay)
* Medical comorbidities that in the opinion of the investigator limits the patient's ability to complete the study
* Symptomatic metastases (Metastases allowed if asymptomatic)
* Current use of appetite suppressant medications
* Current use of any weight loss medications including herbal weight loss supplements or if patients are enrolled in a diet/weight loss program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Mean change in weight | 6 months
  Difference in change in weight between pre- and post- intervention between carbohydrate restricted and control group

SECONDARY OUTCOMES:
Changes in serum estradiol | 6 months
  Difference in changes in serum estradiol between pre- and post-intervention between low-carbohydrate group and control group
Changes in fasting glucose | 6 months
  Difference in changes in fasting glucose between pre- and post-intervention between low-carbohydrate group and control group
Changes in insulin | 6 months
  Difference in changes in insulin between pre- and post-intervention between low-carbohydrate group and control group
Changes in HbA1c | 6 months
  Difference in changes in HbA1c between pre- and post-intervention between low-carbohydrate group and control group
Changes in triglycerides | 6 months
  Difference in changes in triglycerides between pre- and post-intervention between low-carbohydrate group and control group
Changes in LDL | 6 months
  Difference in changes in LDL between pre- and post-intervention between low-carbohydrate group and control group
Changes in HDL | 6 months
  Difference in changes in HDL between pre- and post-intervention between low-carbohydrate group and control group
Changes in cholesterol | 6 months
  Difference in changes in cholesterol between pre- and post-intervention between low-carbohydrate group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Farin Amersi, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No